CLINICAL TRIAL: NCT02539368
Title: POST-MARKETING OBSERVATIONAL COHORT STUDY OF PATIENTS WITH INFLAMMATORY BOWEL DISEASE (IBD) TREATED WITH CT-P13 IN USUAL CLINICAL PRACTICE (CONNECT-IBD)
Brief Title: Post-Marketing Use Of CT-P13 (Infliximab) For Standard Of Care Treatment Of Inflammatory Bowel Disease
Acronym: CONNECT-IBD
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: ZOB INF 1402; C1231001 (Other: Alias Study Number)
Record Dates: First submitted 2015-07-22; First posted 2015-09-03 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn's Disease
Keywords: CT-P13; Inflectra; Remicade; Infliximab; Observational; Follow-up; Safety; Effectiveness
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — CT-P13; Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CT-P13: biosimilar infliximab
  Interventions: Drug: CT-P13
- Remicade: infliximab
  Interventions: Drug: Remicade

INTERVENTIONS:
Drug: CT-P13 — biosimilar infliximab
  Other Names: Inflectra; Remsima
  Groups: CT-P13
Drug: Remicade — infliximab
  Groups: Remicade

SUMMARY:
This is a post-marketing observational study of patients with Inflammatory Bowel Disease (specifically, Crohn's disease or Ulcerative Colitis) who have been prescribed CT-P13 (infliximab) or Remicade (infliximab) for treatment. CT-P13 (brand names Inflectra and Remsima) is a biosimilar medicine to Remicade, meaning it is a biologic medicine that contains the same active substance as Remicade (infliximab). The key study objectives are as follows:

* To characterize the population and drug utilization patterns of patients treated with CT-P13 for Crohn's Disease (CD) or Ulcerative Colitis (UC) in the context of standard of care Remicade
* To explore the long-term safety profile of CT-P13 in the treatment of patients with CD or UC in the context of standard of care Remicade
* To assess the effectiveness of CT-P13 in the treatment of patients with CD or UC in the context of standard of care Remicade

DETAILED DESCRIPTION:
The study will be conducted in accordance with legal and regulatory requirements with scientific purpose, value and rigor following generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP), Good Epidemiological Practice (GEP), Good Practices for Outcomes Research, International Ethical Guidelines for Epidemiological Research, European Medicines Agency (EMA) European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) Guide on Methodological Standards in Pharmacoepidemiology, and FDA Guidance for Industry. Data sources will be validated and will consist of the hospital medical records and monitoring will be organized on a regular basis. Data for the study will be entered into a web based electronic data capture (EDC) system at enrolment and then approximately every 3 months (at a minimum) thereafter up to 2 years. Adverse events will be encoded according to MedDRA 17.1 or later. The sample size will be approximately 2500 patients recruited over a 30 month period and followed up to 2 years. No inferential analyses are planned. Statistical analysis will be descriptive in nature.

ELIGIBILITY:
Inclusion Criteria:

1. At least 12 years of age at the time of initial confirmed diagnosis of CD or UC and at least 18 years of age at the time of enrolment to the study.
2. Patients who are prescribed CT-P13 or Remicade for the treatment of CD or UC prescribed according to the corresponding summary of product characteristics (SmPC) as determined by the Investigator. Patients with stomas or surgery/pouch will be included.

Exclusion Criteria:

1. Any reported contraindications for CT-P13 or Remicade, according to the SmPC.
2. Known hypersensitivity (including severe, acute infusion reactions) to infliximab, its excipients or other murine proteins, at the time of enrolment.
3. Prior history of failure to respond to Remicade or CT-P13.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will include patients with CD or UC, who are being treated, or initiating treatment, with CT-P13 or Remicade at the time of study enrolment. This would include the following treatment subgroups:
  * Biologic-naïve patients initiating CT-P13 (or Remicade);
  * Patients currently being treated with CT-P13 (or Remicade);
  * Patients who are considered stable by the Investigator under Remicade therapy for CD or UC, who switch to CT-P13;
  * Patients switching to CT-P13 or Remicade from an alternative biologic therapy (e.g. adalimumab) due to non-responsiveness to or intolerance;
  * Patients re-initiating CT-P13 or Remicade after having successfully completed and exited a previous course of infliximab therapy in the past.
  * Patients with fistulating disease or stomas and those receiving combination therapy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2565 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (140):
- Belgium (2):
  - UZ Leuven Campus Gasthuisberg, Leuven, Vlaams Brabant
  - UZ Antwerpen, Edegem
- Czechia (5):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Hradecká Poliklinika III, HEPATO-GASTROENTEROLOGIE HK, s.r.o, Hradec Králové
  - Centrum péce o zažívací trakt, Vítkovická nemocnice, Ostrava - Vitkovice
  - IKEM (Institut Klinické a Experimentální Medicíny), Prague
  - Nemocnice Na Bulovce, Praha 8 Liben
- Finland (3):
  - Keski-Suomen keskussairaala, Jyväskylä
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- France (30):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHRU de Besancon, Besançon
  - Centre Hospitalier Universitaire, Caen
  - Clinique de Bercy, Charenton
  - CHU Clermontferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hôpital Louis Mourier, Colombes
  - CHU de Grenoble, Grenoble
  - CHRU, Lille
  - Hopital Edouard Herriot Pav H, Lyon
  - Hopital Europeen, Marseille
  - Hopital Nord, Marseille
  - CHU, Montpellier
  - CHU Nimes, Nîmes
  - Hôpital Saint-Antoine, AP-HP, Universite Pierre-et-Marie-Curie, Paris
  - Hopital Cochin, Paris
  - Institut Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital St Louis, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - Hopital Metz Tessy, Pringy
  - Hopital Robert Debre, Reims
  - Chu Ch.Nicolle, Rouen
  - Service: CHU saint-etienne, Saint Priez En Jarez
  - Centre Hospitalier Universitaire, Strasbourg
  - CHU Rangueil, Toulouse
  - Hopital Purpan, Toulouse
  - CHU Nancy, Vandœuvre-lès-Nancy
  - Groupe hospitalier mutualiste les portes du Sud, Vénissieux
- Germany (25):
  - St. Marienkrankenhaus, Ludwigshafen am Rhein, Gartenstadt
  - Gemeinschaftspraxis im MEDICUM, Altenholz
  - Gastroenterologische Praxis Dr. med. B. Adami, Alzey
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Gastroenterologie Am Bayerischen Platz, Berlin
  - Kreiskliniken Altotting-Burghausen, Burghausen
  - Interdisciplinaeres Crohn-Colitis Centrum Rhein-Main, Frankfurt am Main
  - Gemeinschaftspraxis Dr. R Denger und Dr. T. Pfitzner, Friedrichsthal
  - PraxisZentrum fuer Gastroenterologie, Grevenbroich
  - Hamburgisches Forschungsinstitut fur chronisch entzuendliche, Hamburg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Internisten am Markt Dres. Schwerdtfeger & Lehmann, Köthen
  - Internistische Gemeinschaftspraxis fuer Verdauungs- und Stoffwechselerkrankungen, Leipzig
  - Onco Studies an der Onkologie Dreiländereck, Loerrach
  - Universitaetsmedizin Mannheim, Mannheim
  - Magen-Darm Praxis Prof. Dr. Krammer & Kollegen, Mannheim
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Praxis Prof.Dr. med. Herbert Kellner, Muenchen-Nymphenburg
  - Medizinisches Versorgungszentrum Portal 10, Münster
  - Gastroenterologische Gemeinschaftspraxis am Germania-Campus, Münster
  - Praxiszentrum Alte Maelzerei, Regensburg
  - Magen-Darm-Zentrum Remscheid, Remscheid
  - Zentrum für Gastroenterologie Saarbrücken MVZ GmbH, Saarbrücken
  - Ambulanzzentrum-Schweinfurt, Schweinfurt
  - Gastroenterologische Schwerpunktpraxis Stuttgart, Stuttgart
- Greece (7):
  - University Hospital of Patras, Rio, Patra, Achaia
  - Hippokration General Hospital of Athens, Athens, Attica
  - Venizeleio Hospital of Heraklion, Heraklion, Crete
  - Evangelismos Hospital, Athens
  - University Hospital of Ioannina, Ioannina
  - University Hospital of Larissa, Larissa
  - General Hospital of Thessaloniki Ippokrateio, Thessaloniki
- Hungary (3):
  - Semmelweis University, Budapest
  - MH Egeszsegugyi Kozpont - Honvedkorhaz, Budapest
  - Szte szent-gyorgyi albert klinikai kozpont, Szeged
- Italy (23):
  - Presidio Ospedaliero "M. Raimondi", San Cataldo (Caltanisetta), Caltanisetta
  - ASL 11 Empoli - Ospedale San Giuseppe, Empoli, FI
  - Azienda Ospedaliero Universitaria Careggi, Florence, FI
  - I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milano
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Ospedale "Sacro Cuore - Don Calabria", Negrar, Verona
  - Fondazione Poliambulanza - Istituto Ospedaliero, Brescia
  - Azienda Ospedaliera per l'Emergenza Cannizzaro, Catania
  - Azienda Ospedaliero Universitaria - Policlinico "Vittorio Emanuele", Catania
  - Università degli Studi "G. d'Annunzio" Chieti - Pescara, Chieti
  - ASUR Area Vasta n. 4 - Ospedale A. Murri, Fermo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Università degli Studi di Genova, Genova
  - Ospedale Generale Provinciale di Macerata, Macerata
  - A.O.U. Policlinico "G.Martino", Messina
  - Azienda Ospedaliera - Universitaria di Modena Policlinico, Modena
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Az.Osp. Ospedali Riuniti 'Villa Sofia-Cervello, Palermo
  - AOUP - Ospedale di Cisanello, Pisa
  - Azienda Ospedaliera Universitaria di PISA, Pisa
  - Ospedale Sandro Pertini, Roma
  - Ospedale San Camillo, Rome
  - A.O.U. "S. Maria della Misericordia di Udine", Udine
- Netherlands (3):
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Rijnstate, Gelderland
- Portugal (4):
  - Hospital Prof. Doutor Fernando Fonseca E.P.E, Amadora, Lisbon District
  - Centro Hospitalar entre Douro e Vouga E.P.E., Santa Maria Da Feira, Porto District
  - Centro Hospitalar Barreiro Montijo, E.P.E, Barreiro
  - Centro Hospitalar Lisboa Norte, E.P.E.- Hospital Santa Maria, Lisbon
- Slovakia (2):
  - FNsP F. D. Roosevelta Banska Bystrica, Banská Bystrica
  - V. interna klinika LFUK a UNB, Ambulancia pre nespecificke zapalove ochorenia, Bratislava
- Spain (23):
  - Hospital Arquitecto Marcide, Ferrol, A Coruna
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital Son Espases, Palma. Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Barcelona
  - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital de Galdakao, Usansolo, Bizkaia
  - Hospital Universitario de Gran Canaria DR NEGRIN, Las Palmas de Gran Canari, Canary Islands
  - Hospital de Alcorcon, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Infanta Sofia, San Sebastian de Los Reye, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Alvaro Cunqueiro, Pontevedra
  - Hospital Clínico de Valencia, Valencia
  - Consorci Hospital General Universitari de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (10):
  - Royal Gwent Hospital, Exeter, Devon
  - Dorset County Hospital, Dorchester, Dorset
  - Gloucestershire Hospitals - NHS Foundation Trust, Gloucester, Gloucestershire
  - Cwm Taf University Health Board, Llantrisant, Wales
  - University Hospital Coventry, Coventry, WEST Midlands
  - Salisbury NHS Foundation Trust, Salisbury, Wiltshire
  - Heart of England NHS Foundation Trust, Birmingham
  - The Royal Bournemouth Hospital, Bournemouth
  - Queen Alexandra Hospital, Hampshire
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Bokemeyer B, Hlavaty T, Allez M, Selema P, Moosavi S, Cadatal MJ, Fowler H, Mueller M, Liau KF, Gisbert JP. Real-world observational cohort study of treatment patterns and safety outcomes of infliximab biosimilar CT-P13 for the treatment of inflammatory bowel disease (CONNECT-IBD). Expert Opin Biol Ther. 2023 Jul-Dec;23(8):791-800. doi: 10.1080/14712598.2023.2200883. Epub 2023 Apr 16. PMID 37038897

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2565 participants were enrolled in the study, out of which 22 participants were not eligible to receive treatment for any of the treatment groups. Hence, only those participants who received treatment during the study observation period were included in the participants flow section.
Groups:
- CT-P13: Participants diagnosed with either Crohn's Disease (CD) or Ulcerative Colitis (UC), and who were biologic naive initiating CT-P13 and received CT-P13 continuously, or participants who were treated with CT-P13 continuously, or who were treated with CT-P13 then switched to other anti-tumor necrosis factors (TNFs) therapy except Remicade or non-biologic treatment during the study, or those who switched to CT-P13 from an alternative biologic therapy (except Remicade) due to non-responsiveness to or intolerance with existing therapy were enrolled in this group. Participants received CT-P13 continuously in accordance with usual clinical practice of Inflammatory bowel disease (IBD) at the discretion of the physician and observed for a duration of approximately 24 months.
- Remicade: Participants diagnosed with either CD or UC, and who were biologic naive initiating Remicade and received Remicade continuously, or participants who were treated with Remicade continuously, or who were treated with Remicade then switched to other anti-TNFs therapy (except CT-P13) or non-biologic treatment during the study, or those who switched to Remicade from an alternative biologic therapy (except CT-P13) due to non-responsiveness or intolerance were enrolled in this group. Participants received Remicade in accordance with usual clinical practice of IBD at the discretion of the physician and observed for a duration of approximately 24 months.
- Switched From Remicade to CT-P13: Participants diagnosed with either CD or UC and who were previously treated with Remicade continuously as per usual clinical practice of IBD, switched to CT-P13 once, either at enrollment or during the study were observed for a duration of approximately 24 months.
- Switched From CT-P13 to Remicade: Participants diagnosed with either CD or UC and who were previously treated with CT-P13 continuously as per usual clinical practice of IBD, switched to Remicade once, either at enrollment or during the study were observed for a duration of approximately 24 months.
- Multiple Switchers: Participants with CD or UC with at least 2 switches between Remicade and CT-P13 during the study, were observed for a duration of approximately 24 months. Both Remicade and CT-P13 were administered as per usual clinical practice of IBD.
Period: Overall Study
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Started | 1522 | 494 | 358 | 67 | 102
Completed | 1117 | 393 | 291 | 60 | 88
Not Completed | 405 | 101 | 67 | 7 | 14
Not completed — Death | 4 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 44 | 35 | 9 | 1 | 3
Not completed — Physician Decision | 49 | 15 | 7 | 0 | 2
Not completed — Lost to Follow-up | 96 | 21 | 16 | 4 | 3
Not completed — Adverse Event | 44 | 5 | 9 | 0 | 3
Not completed — Participant Non-compliant | 13 | 2 | 1 | 1 | 0
Not completed — Other | 145 | 18 | 24 | 1 | 3
Not completed — Missing | 10 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study drug during the observation period.
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers | Total
Number analyzed (Participants) | 1522 | 494 | 358 | 67 | 102 | 2543
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (14.65) | 38.8 (12.74) | 40.9 (14.14) | 41.1 (13.96) | 38.4 (13.23) | 39.8 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 750 | 233 | 158 | 29 | 48 | 1218
  Male | 772 | 261 | 200 | 38 | 54 | 1325
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 0 | 0 | 0 | 5
  Asian | 5 | 3 | 5 | 0 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 7 | 0 | 1 | 0 | 0 | 8
  White | 1080 | 391 | 275 | 55 | 83 | 1884
  Other | 267 | 60 | 49 | 11 | 14 | 401
  Unknown or Not Reported | 158 | 39 | 28 | 1 | 5 | 231
Participants With Medical History of Smoking [Count of Participants; unit: Participants] | 320 | 94 | 70 | 12 | 17 | 513
Participants With a History of Cancer [Count of Participants; unit: Participants] | 41 | 10 | 6 | 1 | 4 | 62
Participants With Stoma Status [Count of Participants; unit: Participants] | 33 | 13 | 14 | 3 | 2 | 65
Participants With a History Surgery [Count of Participants; unit: Participants] — Surgery status was a categorical variable defined as yes if the participant had prior surgical treatment related to the treatment of CD or UC.
  Participants | 395 | 165 | 116 | 23 | 32 | 731
Participants With a History of Fistula Disease [Count of Participants; unit: Participants] | 304 | 124 | 86 | 19 | 28 | 561

OUTCOME MEASURES:

1. Primary Outcome: Disease Characteristics of Participants: Disease Duration
Description: Disease duration was defined as the number of months from initial diagnosis of inflammatory bowel disease (CD or UC) to the date of informed consent, which was recorded at the time of enrollment into the study (baseline).
Time Frame: Baseline (Day 1)
Population: Safety analysis population included all participants who received at least 1 dose of study drug during the observation period. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1519 | 494 | 358 | 67 | 102
months | 63.0 [0 to 579] | 112.5 [0 to 632] | 120.0 [2 to 593] | 86.0 [0 to 519] | 101.0 [9 to 457]

2. Primary Outcome: Number of Participants Who Switched Treatment
Description: Here, number of participants with either UC or CD, who switched from remicade to CT-P13; switched from CT-P13 to remicade and multiple switchers were reported.
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 358 | 67 | 102
Participants
  Crohn's Disease | 237 | 47 | 72
  Ulcerative Colitis | 121 | 20 | 30

3. Primary Outcome: Reasons for Switching Treatment by Participants
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: Reasons for switch were not captured in electronic data capture. Hence, due to change in planned analysis, data was not collected and analyzed.
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Total Dose of Infusion Received
Description: Total dose of infusion received by the participants was calculated.
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: milligram
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1520 | 493 | 358 | 67 | 102
milligram | NA [NA to NA] — Due to inconsistency in reporting of total daily dose, the median total dose and full range could not be estimated. | NA [NA to NA] — Due to inconsistency in reporting of total daily dose, the median total dose and full range could not be estimated. | NA [NA to NA] — Due to inconsistency in reporting of total daily dose, the median total dose and full range could not be estimated. | NA [NA to NA] — Due to inconsistency in reporting of total daily dose, the median total dose and full range could not be estimated. | NA [NA to NA] — Due to inconsistency in reporting of total daily dose, the median total dose and full range could not be estimated.

5. Primary Outcome: Number of Participants by Frequency of Infusion Received
Description: Number of participants by infusion frequency (weeks) were reported at baseline and categorized as follows: once a week; once every 2 weeks; once every 3 weeks; once every 4 weeks; once every 5 weeks; once every 6 weeks; once every 7 weeks; once every 8 weeks and others. Here, 'Others' category included all the frequencies apart from the mentioned categories.
Time Frame: Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1283 | 433 | 317 | 60 | 85
Participants
  Once a week | 5 | 0 | 0 | 0 | 0
  Once every 2 weeks | 140 | 5 | 11 | 3 | 3
  Once every 3 weeks | 1 | 0 | 0 | 0 | 1
  Once every 4 weeks | 109 | 47 | 32 | 9 | 7
  Once every 5 weeks | 7 | 8 | 5 | 0 | 4
  Once every 6 weeks | 84 | 67 | 43 | 3 | 15
  Once every 7 weeks | 9 | 27 | 14 | 2 | 4
  Once every 8 weeks | 804 | 247 | 198 | 42 | 47
  Other | 124 | 32 | 14 | 1 | 4

6. Primary Outcome: Number of Participants Who Had Change in Infusion Dose
Description: Participants who had change in the dose of infusion (either dose reduction or increase in dose) were included and reported.
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1522 | 494 | 358 | 67 | 102
Participants | 479 | 110 | 89 | 28 | 31

7. Primary Outcome: Number of Participants Who Had Change in Infusion Dose Categorized Based on Reasons of Change
Description: Participants who had change in infusion dose due to various reasons such as principal investigator's decision, participant's decisions, loss of response, lack of compliance, hypersensitivity, occurrence of adverse event (including adverse event special interest [AESI]/ serious adverse event [SAE]), positive for antibodies and other were reported. Here, 'Others' category included all reasons apart from the mentioned categories. A participant could have different reasons of dose change across visits, hence could be counted in more than one category.
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 479 | 110 | 89 | 28 | 31
Participants
  Principal Investigator's Decision | 213 | 61 | 31 | 26 | 16
  Participant's Decision | 5 | 2 | 0 | 0 | 0
  Loss of response | 142 | 27 | 17 | 3 | 12
  Lack of compliance | 3 | 1 | 0 | 0 | 0
  Hypersensitivity | 4 | 1 | 1 | 0 | 0
  Occurrence of Adverse Event (including AESI/SAE) | 23 | 3 | 3 | 0 | 2
  Positive for antibodies | 5 | 2 | 2 | 0 | 0
  Other | 142 | 26 | 42 | 2 | 9

8. Primary Outcome: Number of Participants Who Took Concomitant Medications Related to the Treatment of Crohn's Disease (CD) or Ulcerative Colitis (UC)
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1522 | 494 | 358 | 67 | 102
Participants | 1025 | 262 | 187 | 39 | 67

9. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Event (AEs), Serious Adverse Events (SAEs) and Adverse Event With Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent were events between first dose of infusion up to month 24, that were absent before treatment or that worsened relative to pretreatment state. Hypersensitivity was the pre-defined TEAE of special Interest for this study. AEs included both serious and non-serious adverse events.
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1522 | 494 | 358 | 67 | 102
Participants
  TEAEs | 621 | 133 | 130 | 15 | 30
  SAEs | 256 | 43 | 57 | 10 | 15
  TEAEs of Special Interest | 189 | 49 | 37 | 8 | 11

10. Secondary Outcome: Number of Participants Remaining in Clinical Remission or Relapse
Description: Clinical remission in participants was defined by a total Mayo score of 2 points or lower, with no individual sub score exceeding 1 point. Mayo score is an instrument designed to measure disease activity. It consisted of 4 sub scores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and physician's global assessment, each sub score graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease. The relapse of clinical remission was defined as the time from the date of first attaining CR to the date of relapse or death from any cause, whichever occurred first.
Time Frame: Months 6, 12, 18 and 24
Population: Full analysis set (FAS)=all participants who received at least 1 dose of study drug and had at least one post-dose assessment of any of the effectiveness outcomes (clinical assessment of disease activity, laboratory and imaging results related to assessment of CD or UC).Number analyzed =participants evaluable at specified time points for each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1516 | 492 | 358 | 67 | 102
Participants
  Month 6: number analyzed (Participants) | 1036 | 335 | 280 | 54 | 74
  Month 6: Remission | 870 | 312 | 261 | 51 | 70
  Month 6: Relapse | 166 | 23 | 19 | 3 | 4
  Month 12: number analyzed (Participants) | 914 | 306 | 240 | 47 | 64
  Month 12: Remission | 802 | 288 | 224 | 45 | 58
  Month 12: Relapse | 112 | 18 | 16 | 2 | 6
  Month 18: number analyzed (Participants) | 703 | 268 | 203 | 32 | 66
  Month 18: Remission | 633 | 257 | 192 | 31 | 61
  Month 18: Relapse | 70 | 11 | 11 | 1 | 5
  Month 24: number analyzed (Participants) | 424 | 191 | 157 | 24 | 43
  Month 24: Remission | 386 | 184 | 148 | 23 | 39
  Month 24: Relapse | 38 | 7 | 9 | 1 | 4

11. Secondary Outcome: Crohn's Disease: Number of Participants With Shift From Baseline in Harvey Bradshaw Index (HBI) According to Clinical Remission
Description: HBI is a simple index of CD activity. HBI measures 5 parameters; the general well-being (ranging from 0=very well to 4=terrible), abdominal pain ranging from 0 (none) to 3 (severe), number of liquid stools per day (no maximum score), presence of an abdominal mass on physical exam ranging from 0 (none) to 3 (definite and tender), and whether there are any complications ranging from 0=no complications, 1=Arthralgia; 2=Uveitis; 3=Erythema nodosum; 4=Aphthous ulcer; 5=Pyoderma gangrenosum; 6=Anal fissure; 7=New fistula and 8=abscess). The total HBI score is the sum of all the 5 individual parameters, the minimum score is 0 and there was no pre-specified maximum score as it depends on the number of liquids stools. Higher HBI scores=greater disease activity. The level of disease activity was interpreted as clinical remission (CR) (score less than [<] 5), mild disease (MD) (score equal to [=] 5 to 7), moderate disease (Mod D) (score=8 to 16) and severe disease (SD) (score more than [>] 16).
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: FAS =all participants who received at least 1 dose of study drug and had at least one post-dose assessment of any of the effectiveness outcomes. Here, Overall number of participants analyzed =Number of participants evaluable for this outcome measure. Number analyzed =participants evaluable at specified time points for each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 969 | 348 | 237 | 47 | 72
Participants
  At Baseline | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 6-CR: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 6-CR | 485 | 211 | 125 | 24 | 43
  Baseline-CR; Month 6-MD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 6-MD | 42 | 11 | 11 | 2 | 4
  Baseline-CR; Month 6-Mod D: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 6-Mod D | 23 | 8 | 2 | 1 | 0
  Baseline-CR; Month 6-SD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 6-SD | 1 | 1 | 0 | 0 | 0
  Baseline-CR; Month 6-Missing: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 6-Missing | 55 | 15 | 12 | 2 | 2
  Baseline-CR; Month 12-CR: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 12-CR | 429 | 182 | 109 | 22 | 42
  Baseline-CR; Month 12-MD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 12-MD | 36 | 14 | 8 | 3 | 1
  Baseline-CR; Month 12-Mod D: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 12-Mod D | 20 | 4 | 5 | 1 | 0
  Baseline-CR; Month 12-SD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 12-SD | 0 | 0 | 0 | 0 | 0
  Baseline-CR; Month 12-Missing: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 12-Missing | 121 | 46 | 28 | 3 | 6
  Baseline-CR; Month 18-CR: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 18-CR | 326 | 143 | 96 | 17 | 37
  Baseline-CR; Month 18-MD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 18-MD | 25 | 11 | 4 | 0 | 1
  Baseline-CR; Month 18-Mod D: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 18-Mod D | 8 | 4 | 2 | 0 | 1
  Baseline-CR; Month 18-SD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 18-SD | 0 | 0 | 0 | 0 | 0
  Baseline-CR; Month 18-Missing: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 18-Missing | 247 | 88 | 48 | 12 | 10
  Baseline-CR; Month 24-CR: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 24-CR | 194 | 98 | 68 | 11 | 28
  Baseline-CR; Month 24-MD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 24-MD | 16 | 7 | 3 | 1 | 2
  Baseline-CR; Month 24-Mod D: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 24-Mod D | 5 | 1 | 3 | 0 | 0
  Baseline-CR; Month 24-SD: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 24-SD | 0 | 0 | 1 | 0 | 0
  Baseline-CR; Month 24-Missing: number analyzed (Participants) | 606 | 246 | 150 | 29 | 49
  Baseline-CR; Month 24-Missing | 391 | 140 | 75 | 17 | 19

12. Secondary Outcome: Crohn's Disease: Number of Participants With Shift From Baseline in Harvey Bradshaw Index According to Disease Activity
Description: HBI is a simple index of CD activity. HBI measures 5 clinical parameters; the general well-being ranging from 0 (very well) to 4 (terrible), abdominal pain ranging from 0 (none) to 3 (severe), number of liquid stools per day (no maximum score), presence of an abdominal mass on physical exam ranging from 0 (none) to 3 (definite and tender), and whether there are any complications ranging from 0=no complications, 1=Arthralgia; 2=Uveitis; 3=Erythema nodosum; 4=Aphthous ulcer; 5=Pyoderma gangrenosum; 6=Anal fissure; 7=New fistula and 8=abscess). The total HBI score is the sum of all the 5 individual parameters, the minimum score is 0 and there was no pre-specified maximum score as it depends on the number of liquids stools. Higher HBI scores=greater disease activity. The level of disease activity was interpreted as clinical remission (CR) (HBI score < 5), mild disease (MD) (HBI score = 5 to 7), moderate disease (Mod D) (HBI score = 8 to 16) and severe disease (SD) (HBI score >16).
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 969 | 348 | 237 | 47 | 72
Participants
  At Baseline: MD | 137 | 45 | 24 | 10 | 7
  At Baseline: Mod D | 91 | 22 | 15 | 4 | 3
  At Baseline: SD | 6 | 2 | 0 | 0 | 0
  Baseline-MD; Month 6-CR: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 6-CR | 82 | 21 | 9 | 5 | 3
  Baseline-MD; Month 6-MD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 6-MD | 30 | 13 | 11 | 4 | 1
  Baseline-MD; Month 6-Mod D: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 6-Mod D | 12 | 8 | 3 | 0 | 2
  Baseline-MD; Month 6-SD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 6-SD | 0 | 0 | 1 | 0 | 1
  Baseline-MD; Month 6-Missing: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 6-Missing | 13 | 3 | 0 | 1 | 0
  Baseline-Mod D; Month 6-CR: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 6-CR | 39 | 4 | 6 | 3 | 2
  Baseline-Mod D; Month 6-MD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 6-MD | 19 | 6 | 2 | 1 | 0
  Baseline-Mod D; Month 6-Mod D: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 6-Mod D | 25 | 8 | 6 | 0 | 0
  Baseline-Mod D; Month 6-SD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 6-SD | 1 | 0 | 0 | 0 | 0
  Baseline-Mod D; Month 6-Missing: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 6-Missing | 7 | 4 | 1 | 0 | 1
  Baseline-SD; Month 6-CR: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 6-CR | 1 | 1 | 0 | 0 | 0
  Baseline-SD; Month 6-MD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 6-MD | 2 | 0 | 0 | 0 | 0
  Baseline-SD; Month 6-Mod D: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 6-Mod D | 2 | 0 | 0 | 0 | 0
  Baseline-SD; Month 6-SD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 6-SD | 0 | 1 | 0 | 0 | 0
  Baseline-SD; Month 6-Missing: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 6-Missing | 1 | 0 | 0 | 0 | 0
  Baseline-MD; Month 12-CR: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 12-CR | 81 | 24 | 14 | 6 | 4
  Baseline-MD; Month 12-MD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 12-MD | 16 | 6 | 3 | 2 | 1
  Baseline-MD; Month 12-Mod D: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 12-Mod D | 7 | 6 | 3 | 0 | 1
  Baseline-MD; Month 12-SD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 12-SD | 1 | 0 | 0 | 0 | 1
  Baseline-MD; Month 12-Missing: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 12-Missing | 32 | 9 | 4 | 2 | 0
  Baseline-Mod D; Month 12-CR: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 12-CR | 39 | 6 | 4 | 3 | 3
  Baseline-Mod D; Month 12-MD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 12-MD | 15 | 9 | 0 | 1 | 0
  Baseline-Mod D; Month 12-Mod D: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 12-Mod D | 16 | 2 | 6 | 0 | 0
  Baseline-Mod D; Month 12-SD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 12-SD | 0 | 0 | 0 | 0 | 0
  Baseline-Mod D; Month 12-Missing: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 12-Missing | 21 | 5 | 5 | 0 | 0
  Baseline-SD; Month 12-CR: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 12-CR | 1 | 1 | 0 | 0 | 0
  Baseline-SD; Month 12-MD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 12-MD | 2 | 0 | 0 | 0 | 0
  Baseline-SD; Month 12-Mod D: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 12-Mod D | 1 | 0 | 0 | 0 | 0
  Baseline-SD; Month 12-SD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 12-SD | 0 | 1 | 0 | 0 | 0
  Baseline-SD; Month 12-Missing: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 12-Missing | 2 | 0 | 0 | 0 | 0
  Baseline-MD; Month 18-CR: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 18-CR | 60 | 24 | 12 | 2 | 2
  Baseline-MD; Month 18-MD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 18-MD | 10 | 6 | 1 | 4 | 3
  Baseline-MD; Month 18-Mod D: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 18-Mod D | 4 | 2 | 1 | 0 | 2
  Baseline-MD; Month 18-SD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 18-SD | 2 | 0 | 0 | 0 | 0
  Baseline-MD; Month 18-Missing: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 18-Missing | 61 | 13 | 10 | 4 | 0
  Baseline-Mod D; Month 18-CR: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 18-CR | 30 | 4 | 2 | 3 | 2
  Baseline-Mod D; Month 18-MD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 18-MD | 13 | 7 | 2 | 1 | 1
  Baseline-Mod D; Month 18-Mod D: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 18-Mod D | 14 | 3 | 3 | 0 | 0
  Baseline-Mod D; Month 18-SD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 18-SD | 0 | 0 | 0 | 0 | 0
  Baseline-Mod D; Month 18-Missing: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 18-Missing | 34 | 8 | 8 | 0 | 0
  Baseline-SD; Month 18-CR: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 18-CR | 1 | 1 | 0 | 0 | 0
  Baseline-SD; Month 18-MD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 18-MD | 2 | 1 | 0 | 0 | 0
  Baseline-SD; Month 18-Mod D: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 18-Mod D | 1 | 0 | 0 | 0 | 0
  Baseline-SD; Month 18-SD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 18-SD | 0 | 0 | 0 | 0 | 0
  Baseline-SD; Month 18-Missing: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 18-Missing | 2 | 0 | 0 | 0 | 0
  Baseline-MD; Month 24-CR: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 24-CR | 34 | 13 | 8 | 5 | 2
  Baseline-MD; Month 24-MD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 24-MD | 15 | 6 | 2 | 1 | 2
  Baseline-MD; Month 24-Mod D: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 24-Mod D | 2 | 1 | 1 | 0 | 2
  Baseline-MD; Month 24-SD: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 24-SD | 1 | 0 | 0 | 0 | 0
  Baseline-MD; Month 24-Missing: number analyzed (Participants) | 137 | 45 | 24 | 10 | 7
  Baseline-MD; Month 24-Missing | 85 | 25 | 13 | 4 | 1
  Baseline-Mod D; Month 24-CR: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 24-CR | 23 | 3 | 4 | 3 | 1
  Baseline-Mod D; Month 24-MD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 24-MD | 5 | 2 | 1 | 0 | 1
  Baseline-Mod D; Month 24-Mod D: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 24-Mod D | 10 | 9 | 3 | 1 | 0
  Baseline-Mod D; Month 24-SD: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 24-SD | 1 | 0 | 0 | 0 | 0
  Baseline-Mod D; Month 24-Missing: number analyzed (Participants) | 91 | 22 | 15 | 4 | 3
  Baseline-Mod D; Month 24-Missing | 52 | 8 | 7 | 0 | 1
  Baseline-SD; Month 24-CR: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 24-CR | 0 | 1 | 0 | 0 | 0
  Baseline-SD; Month 24-MD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 24-MD | 2 | 0 | 0 | 0 | 0
  Baseline-SD; Month 24-Mod D: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 24-Mod D | 0 | 0 | 0 | 0 | 0
  Baseline-SD; Month 24-SD: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 24-SD | 0 | 1 | 0 | 0 | 0
  Baseline-SD; Month 24-Missing: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0
  Baseline-SD; Month 24-Missing | 4 | 0 | 0 | 0 | 0

13. Secondary Outcome: Ulcerative Colitis: Number of Participants With Shift From Baseline in Partial Mayo Scoring System According to Clinical Remission
Description: Mayo Score is an instrument to measure disease activity of UC. Score ranges from 0 to 12 points. It consists of 4 sub scores, each graded from 0 to 3. Higher scores = more severe disease. A Partial Mayo Score (PMS) (Mayo score without endoscopy) is comprised of 3 parameters: stool frequency ranging from 0 (normal number of stools) to 3 (having >=5 stools more than normal), the presence of rectal bleeding (ranging from 0=no blood seen to 3=blood alone passes), and physician's global assessment (ranging from 0=normal to 3=severe disease). The total partial Mayo score was the sum of all the parameters, score ranging from 0 (normal or inactive disease) to 9 (severe disease). Higher scores indicated more severe disease. The score was calculated if data were available for at least 1 of 3 Mayo sub scores. The level of disease activity was interpreted as clinical remission (CR) (PMS <2), mild disease (MD) (PMS=2 to 4), moderate disease (Mod D) (PMS=5 to 6) and severe disease (SD) (PMS >6).
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 547 | 144 | 121 | 20 | 30
Participants
  At Baseline | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 6-CR: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 6-CR | 117 | 65 | 40 | 7 | 9
  Baseline-CR; Month 6-MD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 6-MD | 27 | 9 | 7 | 2 | 2
  Baseline-CR; Month 6-Mod D: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 6-Mod D | 7 | 0 | 1 | 0 | 1
  Baseline-CR; Month 6-SD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 6-SD | 1 | 0 | 1 | 0 | 0
  Baseline-CR; Month 6-Missing: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 6-Missing | 17 | 9 | 6 | 0 | 1
  Baseline-CR; Month 12-CR: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 12-CR | 107 | 65 | 30 | 8 | 8
  Baseline-CR; Month 12-MD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 12-MD | 24 | 4 | 10 | 0 | 4
  Baseline-CR; Month 12-Mod D: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 12-Mod D | 5 | 0 | 1 | 0 | 1
  Baseline-CR; Month 12-SD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 12-SD | 1 | 0 | 0 | 0 | 0
  Baseline-CR; Month 12-Missing: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 12-Missing | 32 | 14 | 14 | 1 | 0
  Baseline-CR; Month 18-CR: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 18-CR | 88 | 55 | 25 | 3 | 9
  Baseline-CR; Month 18-MD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 18-MD | 13 | 8 | 4 | 0 | 0
  Baseline-CR; Month 18-Mod D: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 18-Mod D | 6 | 0 | 2 | 0 | 3
  Baseline-CR; Month 18-SD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 18-SD | 2 | 0 | 1 | 0 | 0
  Baseline-CR; Month 18-Missing: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 18-Missing | 60 | 20 | 23 | 6 | 1
  Baseline-CR; Month 24-CR: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 24-CR | 57 | 38 | 22 | 3 | 6
  Baseline-CR; Month 24-MD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 24-MD | 7 | 5 | 3 | 0 | 0
  Baseline-CR; Month 24-Mod D: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 24-Mod D | 2 | 1 | 1 | 0 | 0
  Baseline-CR; Month 24-SD: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 24-SD | 0 | 0 | 0 | 0 | 0
  Baseline-CR; Month 24-Missing: number analyzed (Participants) | 169 | 83 | 55 | 9 | 13
  Baseline-CR; Month 24-Missing | 103 | 39 | 29 | 6 | 7

14. Secondary Outcome: Ulcerative Colitis: Number of Participants With Shift From Baseline in Partial Mayo Scoring System According to Disease Activity
Description: Mayo Score is an instrument to measure disease activity of UC. Score ranges from 0 to 12 points. It consists of 4 sub scores, each graded from 0 to 3. Higher scores= more severe disease. A Partial Mayo Score (PMS) (Mayo score without endoscopy) is comprised of 3 parameters: stool frequency ranging from 0 (normal number of stools) to 3 (having >=5 stools more than normal), the presence of rectal bleeding ranging from 0 (no blood seen) to 3 (blood alone passes), and physician's global assessment ranging from 0 (normal) to 3 (severe disease). The total partial Mayo score was the sum of all the parameters, score ranging from 0 (normal or inactive disease) to 9 (severe disease). Higher scores indicated more severe disease. The score was calculated if data were available for at least 1 of 3 Mayo sub scores. The level of disease activity was interpreted as clinical remission (CR) (PMS <2), mild disease (MD) (PMS=2 to 4), moderate disease (Mod D) (PMS=5 to 6) and severe disease (SD) (PMS >6).
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 547 | 144 | 121 | 20 | 30
Participants
  At Baseline: MD | 157 | 30 | 28 | 4 | 9
  At Baseline: Mod D | 76 | 13 | 9 | 3 | 4
  At Baseline: SD | 47 | 5 | 3 | 0 | 1
  Baseline-MD; Month 6-CR: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 6-CR | 71 | 12 | 19 | 3 | 3
  Baseline-MD; Month 6-MD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 6-MD | 48 | 12 | 4 | 1 | 6
  Baseline-MD; Month 6-Mod D: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 6-Mod D | 18 | 2 | 1 | 0 | 0
  Baseline-MD; Month 6-SD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 6-SD | 7 | 0 | 1 | 0 | 0
  Baseline-MD; Month 6-Missing: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 6-Missing | 13 | 4 | 3 | 0 | 0
  Baseline-Mod D; Month 6-CR: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 6-CR | 18 | 3 | 2 | 3 | 2
  Baseline-Mod D; Month 6-MD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 6-MD | 22 | 8 | 5 | 0 | 2
  Baseline-Mod D; Month 6-Mod D: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 6-Mod D | 21 | 0 | 1 | 0 | 0
  Baseline-Mod D; Month 6-SD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 6-SD | 8 | 1 | 0 | 0 | 0
  Baseline-Mod D; Month 6-Missing: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 6-Missing | 7 | 1 | 1 | 0 | 0
  Baseline-SD; Month 6-CR: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 6-CR | 8 | 2 | 0 | 0 | 1
  Baseline-SD; Month 6-MD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 6-MD | 19 | 1 | 1 | 0 | 0
  Baseline-SD; Month 6-Mod D: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 6-Mod D | 6 | 0 | 1 | 0 | 0
  Baseline-SD; Month 6-SD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 6-SD | 7 | 0 | 1 | 0 | 0
  Baseline-SD; Month 6-Missing: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 6-Missing | 7 | 2 | 0 | 0 | 0
  Baseline-MD; Month 12-CR: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 12-CR | 73 | 16 | 14 | 2 | 2
  Baseline-MD; Month 12-MD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 12-MD | 38 | 6 | 7 | 1 | 5
  Baseline-MD; Month 12-Mod D: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 12-Mod D | 10 | 3 | 1 | 0 | 1
  Baseline-MD; Month 12-SD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 12-SD | 3 | 0 | 1 | 1 | 0
  Baseline-MD; Month 12-Missing: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 12-Missing | 33 | 5 | 5 | 0 | 1
  Baseline-Mod D; Month 12-CR: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 12-CR | 24 | 2 | 4 | 2 | 1
  Baseline-Mod D; Month 12-MD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 12-MD | 17 | 6 | 2 | 0 | 2
  Baseline-Mod D; Month 12-Mod D: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 12-Mod D | 6 | 1 | 0 | 0 | 0
  Baseline-Mod D; Month 12-SD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 12-SD | 2 | 0 | 0 | 0 | 0
  Baseline-Mod D; Month 12-Missing: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 12-Missing | 27 | 4 | 3 | 1 | 1
  Baseline-SD; Month 12-CR: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 12-CR | 15 | 2 | 0 | 0 | 1
  Baseline-SD; Month 12-MD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 12-MD | 8 | 1 | 1 | 0 | 0
  Baseline-SD; Month 12-Mod D: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 12-Mod D | 5 | 0 | 2 | 0 | 0
  Baseline-SD; Month 12-SD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 12-SD | 2 | 0 | 0 | 0 | 0
  Baseline-SD; Month 12-Missing: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 12-Missing | 17 | 2 | 0 | 0 | 0
  Baseline-MD; Month 18-CR: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 18-CR | 57 | 14 | 15 | 3 | 3
  Baseline-MD; Month 18-MD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 18-MD | 22 | 5 | 6 | 0 | 2
  Baseline-MD; Month 18-Mod D: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 18-Mod D | 8 | 1 | 1 | 0 | 1
  Baseline-MD; Month 18-SD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 18-SD | 2 | 0 | 0 | 0 | 0
  Baseline-MD; Month 18-Missing: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 18-Missing | 68 | 10 | 6 | 1 | 3
  Baseline-Mod D; Month 18-CR: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 18-CR | 23 | 4 | 2 | 1 | 1
  Baseline-Mod D; Month 18-MD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 18-MD | 16 | 2 | 1 | 0 | 2
  Baseline-Mod D; Month 18-Mod D: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 18-Mod D | 2 | 1 | 1 | 0 | 0
  Baseline-Mod D; Month 18-SD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 18-SD | 0 | 0 | 0 | 0 | 0
  Baseline-Mod D; Month 18-Missing: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 18-Missing | 35 | 6 | 5 | 2 | 1
  Baseline-SD; Month 18-CR: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 18-CR | 15 | 2 | 1 | 0 | 1
  Baseline-SD; Month 18-MD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 18-MD | 5 | 1 | 2 | 0 | 0
  Baseline-SD; Month 18-Mod D: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 18-Mod D | 3 | 0 | 0 | 0 | 0
  Baseline-SD; Month 18-SD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 18-SD | 0 | 0 | 0 | 0 | 0
  Baseline-SD; Month 18-Missing: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 18-Missing | 24 | 2 | 0 | 0 | 0
  Baseline-MD; Month 24-CR: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 24-CR | 43 | 13 | 13 | 2 | 5
  Baseline-MD; Month 24-MD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 24-MD | 10 | 4 | 3 | 0 | 1
  Baseline-MD; Month 24-Mod D: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 24-Mod D | 5 | 1 | 1 | 0 | 0
  Baseline-MD; Month 24-SD: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 24-SD | 0 | 0 | 0 | 0 | 0
  Baseline-MD; Month 24-Missing: number analyzed (Participants) | 157 | 30 | 28 | 4 | 9
  Baseline-MD; Month 24-Missing | 99 | 12 | 11 | 2 | 3
  Baseline-Mod D; Month 24-CR: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 24-CR | 15 | 2 | 0 | 0 | 2
  Baseline-Mod D; Month 24-MD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 24-MD | 11 | 3 | 0 | 0 | 1
  Baseline-Mod D; Month 24-Mod D: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 24-Mod D | 1 | 0 | 1 | 0 | 0
  Baseline-Mod D; Month 24-SD: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 24-SD | 2 | 1 | 1 | 0 | 0
  Baseline-Mod D; Month 24-Missing: number analyzed (Participants) | 76 | 13 | 9 | 3 | 4
  Baseline-Mod D; Month 24-Missing | 47 | 7 | 7 | 3 | 1
  Baseline-SD; Month 24-CR: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 24-CR | 8 | 2 | 0 | 0 | 0
  Baseline-SD; Month 24-MD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 24-MD | 8 | 1 | 1 | 0 | 0
  Baseline-SD; Month 24-Mod D: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 24-Mod D | 1 | 0 | 0 | 0 | 0
  Baseline-SD; Month 24-SD: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 24-SD | 0 | 0 | 0 | 0 | 0
  Baseline-SD; Month 24-Missing: number analyzed (Participants) | 47 | 5 | 3 | 0 | 1
  Baseline-SD; Month 24-Missing | 30 | 2 | 2 | 0 | 1

15. Secondary Outcome: Crohn's Disease: Number of Participants Categorized on the Basis of Montreal Classification Index by Age at Diagnosis
Description: The Montreal classification index for CD was used to classify the extent of the disease activity. It consisted of three parameters: age at diagnosis, location and behavior of the disease activity. There were four different age groups categorized: 16 years or younger, 17-40 years, over 40 years and missing.
Time Frame: At Baseline
Population: FAS =all participants who received at least 1 dose of study drug and had at least one post-dose assessment of any of the effectiveness outcomes. Here, Overall number of participants analyzed =Number of participants evaluable for this outcome measure. Number analyzed =participants evaluable at specified rows for each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 777 | 240 | 164 | 37 | 50
Participants
  16 years or younger | 61 | 33 | 21 | 4 | 6
  17-40 years | 553 | 174 | 115 | 25 | 39
  Over 40 years | 162 | 33 | 28 | 8 | 5
  Missing | 1 | 0 | 0 | 0 | 0

16. Secondary Outcome: Crohn's Disease: Number of Participants Categorized on the Basis of Montreal Classification Index by Location
Description: The Montreal classification index for CD was used to classify the extent of the disease activity. It consisted of three parameters: age at diagnosis, location and behavior of the disease activity. There are four different disease locations presented: Location 1 (L1) is terminal ileum, Location 2 (L2) is colon, Location 3 (L3) is ileocolon and Location 4 (L4) is upper gastrointestinal (GI). The first three categories (L1-L3) was combined with L4 where disease sites coexisted.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 969 | 348 | 237 | 47 | 72
Participants
  At Baseline: Location: number analyzed (Participants) | 777 | 240 | 164 | 37 | 50
  At Baseline: Location: L1 Terminal ileum | 257 | 62 | 34 | 6 | 11
  At Baseline: Location: L2 Colon | 135 | 54 | 32 | 14 | 8
  At Baseline: Location: L3 Ileocolon | 329 | 107 | 80 | 16 | 28
  At Baseline: Location: L4 Upper GI | 14 | 4 | 4 | 1 | 0
  At Baseline: Location: L1 Terminal ileum, L4 Upper GI | 21 | 2 | 1 | 0 | 1
  At Baseline: Location: L2 Colon, L4 Upper GI | 6 | 2 | 1 | 0 | 1
  At Baseline: Location: L3 Ileocolon, L4 Upper GI | 14 | 8 | 12 | 0 | 1
  At Baseline: Location: Missing | 1 | 1 | 0 | 0 | 0
  Month 6: Location: number analyzed (Participants) | 589 | 202 | 127 | 33 | 44
  Month 6: Location: L1 Terminal ileum | 202 | 49 | 26 | 7 | 9
  Month 6: Location: L2 Colon | 105 | 47 | 25 | 12 | 11
  Month 6: Location: L3 Ileocolon | 236 | 94 | 65 | 13 | 22
  Month 6: Location: L4 Upper GI | 12 | 2 | 3 | 1 | 0
  Month 6: Location: L1 Terminal ileum, L4 Upper GI | 15 | 2 | 1 | 0 | 0
  Month 6: Location: L2 Colon, L4 Upper GI | 3 | 3 | 0 | 0 | 0
  Month 6: Location: L3 Ileocolon, L4 Upper GI | 11 | 5 | 7 | 0 | 2
  Month 6: Location: Missing | 5 | 0 | 0 | 0 | 0
  Month 12: Location: number analyzed (Participants) | 468 | 160 | 104 | 33 | 40
  Month 12: Location: L1 Terminal ileum | 150 | 38 | 22 | 7 | 7
  Month 12: Location: L2 Colon | 84 | 40 | 20 | 14 | 10
  Month 12: Location: L3 Ileocolon | 200 | 71 | 55 | 11 | 21
  Month 12: Location: L4 Upper GI | 10 | 3 | 2 | 1 | 1
  Month 12: Location: L1 Terminal ileum, L4 Upper GI | 11 | 2 | 1 | 0 | 0
  Month 12: Location: L2 Colon, L4 Upper GI | 2 | 1 | 0 | 0 | 0
  Month 12: Location: L3 Ileocolon, L4 Upper GI | 8 | 5 | 4 | 0 | 1
  Month 12: Location: Missing | 3 | 0 | 0 | 0 | 0
  Month 18: Location: number analyzed (Participants) | 330 | 124 | 85 | 22 | 36
  Month 18: Location: L1 Terminal ileum | 99 | 28 | 16 | 2 | 8
  Month 18: Location: L2 Colon | 53 | 31 | 18 | 10 | 9
  Month 18: Location: L3 Ileocolon | 150 | 55 | 40 | 8 | 17
  Month 18: Location: L4 Upper GI | 8 | 5 | 4 | 1 | 1
  Month 18: Location: L1 Terminal ileum, L4 Upper GI | 13 | 0 | 0 | 0 | 0
  Month 18: Location: L2 Colon, L4 Upper GI | 2 | 1 | 0 | 0 | 0
  Month 18: Location: L3 Ileocolon, L4 Upper GI | 5 | 4 | 7 | 1 | 1
  Month 18: Location: Missing | 0 | 0 | 0 | 0 | 0
  Month 24: Location: number analyzed (Participants) | 190 | 75 | 57 | 18 | 27
  Month 24: Location: L1 Terminal ileum | 60 | 17 | 15 | 0 | 5
  Month 24: Location: L2 Colon | 41 | 16 | 14 | 9 | 5
  Month 24: Location: L3 Ileocolon | 74 | 33 | 22 | 9 | 14
  Month 24: Location: L4 Upper GI | 7 | 6 | 3 | 0 | 1
  Month 24: Location: L1 Terminal ileum, L4 Upper GI | 2 | 0 | 0 | 0 | 0
  Month 24: Location: L2 Colon, L4 Upper GI | 0 | 1 | 0 | 0 | 0
  Month 24: Location: L3 Ileocolon, L4 Upper GI | 5 | 2 | 3 | 0 | 2
  Month 24: Location: Missing | 1 | 0 | 0 | 0 | 0

17. Secondary Outcome: Crohn's Disease: Number of Participants Categorized on the Basis of Montreal Classification Index by Behavior of the Disease Activity
Description: The Montreal classification index for CD was used to classify the extent of the disease activity. It consists of two parameters: location and behavior of the disease activity. There were 4 different categories for the behavior of the disease activity: Behaviour 1 (B1) was nonstricturing (NS), nonpenetrating (NP); Behaviour 2 (B2) was structuring; Behaviour 3 (B3) was penetrating and p as perianal disease (p). The first 3 categories (B1 to B3) could be added with p to indicate coexisting perianal disease. Perianal disease (p) was defined as the presence of perianal abscesses or fistulae.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 969 | 348 | 237 | 47 | 72
Participants
  At Baseline: Behavior: number analyzed (Participants) | 777 | 240 | 164 | 37 | 50
  At Baseline: Behavior: B1 NS, NP | 324 | 92 | 66 | 9 | 17
  At Baseline: Behavior: B2 Stricturing | 165 | 40 | 43 | 9 | 13
  At Baseline: Behavior: B3 Penetrating | 84 | 32 | 16 | 6 | 6
  At Baseline: Behavior: p Perianal disease | 34 | 5 | 7 | 2 | 3
  At Baseline: Behavior: B2 Stricturing, B3 Penetrating | 1 | 0 | 0 | 0 | 0
  At Baseline: Behavior: B1 NS,NP, p Perianal disease | 77 | 33 | 16 | 5 | 5
  At Baseline: Behavior: B2 Stricturing, p Perianal disease | 32 | 8 | 4 | 1 | 1
  At Baseline: Behavior: B2 Stricturing, B3 Penetrating, p Perianal disease | 0 | 0 | 0 | 0 | 0
  At Baseline: Behavior: B3 Penetrating, p Perianal disease | 57 | 30 | 12 | 5 | 5
  At Baseline: Behavior: Missing | 3 | 0 | 0 | 0 | 0
  Month 6: Behavior: number analyzed (Participants) | 589 | 202 | 127 | 33 | 44
  Month 6: Behavior: B1 NS, NP | 242 | 68 | 46 | 10 | 14
  Month 6: Behavior: B2 Stricturing | 122 | 29 | 36 | 8 | 12
  Month 6: Behavior: B3 Penetrating | 64 | 32 | 14 | 5 | 5
  Month 6: Behavior: p Perianal disease | 27 | 5 | 4 | 1 | 1
  Month 6: Behavior: B2 Stricturing, B3 Penetrating | 0 | 0 | 0 | 0 | 0
  Month 6: Behavior: B1 NS,NP, p Perianal disease | 64 | 34 | 11 | 5 | 6
  Month 6: Behavior: B2 Stricturing, p Perianal disease | 22 | 5 | 3 | 1 | 0
  Month 6: Behavior: B2 Stricturing, B3 Penetrating, p Perianal disease | 1 | 0 | 0 | 0 | 0
  Month 6: Behavior: B3 Penetrating, p Perianal disease | 42 | 29 | 13 | 3 | 6
  Month 6: Behavior: Missing | 5 | 0 | 0 | 0 | 0
  Month 12: Behavior: number analyzed (Participants) | 468 | 160 | 104 | 33 | 40
  Month 12: Behavior: B1 NS, NP | 191 | 56 | 40 | 10 | 17
  Month 12: Behavior: B2 Stricturing | 94 | 26 | 28 | 6 | 9
  Month 12: Behavior: B3 Penetrating | 48 | 26 | 12 | 5 | 2
  Month 12: Behavior: p Perianal disease | 17 | 7 | 1 | 1 | 1
  Month 12: Behavior: B2 Stricturing, B3 Penetrating | 0 | 0 | 0 | 0 | 0
  Month 12: Behavior: B1 NS,NP, p Perianal disease | 60 | 20 | 9 | 6 | 6
  Month 12: Behavior: B2 Stricturing, p Perianal disease | 22 | 5 | 3 | 2 | 0
  Month 12: Behavior: B2 Stricturing, B3 Penetrating, p Perianal disease | 0 | 0 | 0 | 0 | 0
  Month 12: Behavior: B3 Penetrating, p Perianal disease | 33 | 20 | 11 | 3 | 5
  Month 12: Behavior: Missing | 3 | 0 | 0 | 0 | 0
  Month 18: Behavior: number analyzed (Participants) | 330 | 124 | 85 | 22 | 36
  Month 18: Behavior: B1 NS, NP | 135 | 44 | 26 | 4 | 13
  Month 18: Behavior: B2 Stricturing | 77 | 24 | 26 | 4 | 10
  Month 18: Behavior: B3 Penetrating | 26 | 16 | 9 | 4 | 2
  Month 18: Behavior: p Perianal disease | 10 | 4 | 1 | 1 | 0
  Month 18: Behavior: B2 Stricturing, B3 Penetrating | 1 | 0 | 0 | 0 | 0
  Month 18: Behavior: B1 NS,NP, p Perianal disease | 40 | 15 | 11 | 5 | 6
  Month 18: Behavior: B2 Stricturing, p Perianal disease | 14 | 1 | 1 | 0 | 0
  Month 18: Behavior: B2 Stricturing, B3 Penetrating, p Perianal disease | 0 | 0 | 0 | 0 | 0
  Month 18: Behavior: B3 Penetrating, p Perianal disease | 27 | 20 | 11 | 4 | 5
  Month 18: Behavior: Missing | 0 | 0 | 0 | 0 | 0
  Month 24: Behavior: number analyzed (Participants) | 190 | 75 | 57 | 18 | 27
  Month 24: Behavior: B1 NS, NP | 77 | 35 | 20 | 3 | 7
  Month 24: Behavior: B2 Stricturing | 47 | 8 | 15 | 3 | 9
  Month 24: Behavior: B3 Penetrating | 18 | 8 | 4 | 4 | 2
  Month 24: Behavior: p Perianal disease | 4 | 3 | 1 | 1 | 0
  Month 24: Behavior: B2 Stricturing, B3 Penetrating | 0 | 0 | 0 | 0 | 0
  Month 24: Behavior: B1 NS,NP, p Perianal disease | 23 | 8 | 6 | 5 | 5
  Month 24: Behavior: B2 Stricturing, p Perianal disease | 5 | 1 | 1 | 0 | 0
  Month 24: Behavior: B2 Stricturing, B3 Penetrating, p Perianal disease | 0 | 0 | 0 | 0 | 0
  Month 24: Behavior: B3 Penetrating, p Perianal disease | 15 | 12 | 10 | 2 | 4
  Month 24: Behavior: Missing | 1 | 0 | 0 | 0 | 0

18. Secondary Outcome: Ulcerative Colitis: Number of Participants Categorized on the Basis of Montreal Classification Index by Extent
Description: The Montreal classification index for Ulcerative Colitis (UC) was used to classify the extent and severity of the disease activity. There were three subgroups of UC defined by extent: Extent 1 (E1) =Ulcerative proctitis, Extent 2 (E2) =Left-sided UC and Extent 3 (E3) =Extensive UC.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 547 | 144 | 121 | 20 | 30
Participants
  Baseline: number analyzed (Participants) | 380 | 86 | 66 | 16 | 22
  Baseline: E1 Ulcerative proctitis | 41 | 10 | 5 | 0 | 2
  Baseline: E2 Left-sided UC | 151 | 26 | 30 | 3 | 8
  Baseline: E3 Extensive UC | 188 | 50 | 31 | 13 | 12
  Baseline: Missing | 0 | 0 | 0 | 0 | 0
  Month 6: number analyzed (Participants) | 302 | 72 | 50 | 15 | 20
  Month 6: E1 Ulcerative proctitis | 31 | 9 | 1 | 0 | 1
  Month 6: E2 Left-sided UC | 109 | 23 | 24 | 3 | 6
  Month 6: E3 Extensive UC | 159 | 40 | 25 | 12 | 13
  Month 6: Missing | 3 | 0 | 0 | 0 | 0
  Month 12: number analyzed (Participants) | 224 | 66 | 38 | 14 | 18
  Month 12: E1 Ulcerative proctitis | 17 | 7 | 4 | 0 | 1
  Month 12: E2 Left-sided UC | 76 | 21 | 13 | 3 | 7
  Month 12: E3 Extensive UC | 128 | 37 | 21 | 11 | 10
  Month 12: Missing | 3 | 1 | 0 | 0 | 0
  Month 18: number analyzed (Participants) | 168 | 53 | 32 | 8 | 17
  Month 18: E1 Ulcerative proctitis | 15 | 7 | 2 | 0 | 2
  Month 18: E2 Left-sided UC | 55 | 16 | 12 | 1 | 5
  Month 18: E3 Extensive UC | 96 | 29 | 18 | 7 | 10
  Month 18: Missing | 2 | 1 | 0 | 0 | 0
  Month 24: number analyzed (Participants) | 101 | 30 | 25 | 5 | 11
  Month 24: E1 Ulcerative proctitis | 14 | 5 | 2 | 0 | 0
  Month 24: E2 Left-sided UC | 26 | 10 | 8 | 1 | 2
  Month 24: E3 Extensive UC | 59 | 15 | 15 | 4 | 9
  Month 24: Missing | 2 | 0 | 0 | 0 | 0

19. Secondary Outcome: Ulcerative Colitis: Number of Participants Categorized on the Basis of Montreal Classification Index by Severity
Description: The Montreal classification index for UC was used to classify the extent and severity of the disease activity. UC can be classified broadly into four disease activity/severity categories: Severity 0 (S0) = asymptomatic clinical remission; Severity 1 (S1) = Mild UC (passage of four or fewer stools/day [with or without blood], absence of any systemic illness, and normal inflammatory markers); Severity 2 (S2) = Moderate UC (passage of more than four stools per day but with minimal signs of systemic toxicity) and Severity 3 (S3) = Severe UC (passage of at least six bloody stools daily).
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 547 | 144 | 121 | 20 | 30
Participants
  Baseline: number analyzed (Participants) | 380 | 86 | 66 | 16 | 22
  Baseline: S0 | 80 | 46 | 24 | 6 | 6
  Baseline: S1 | 75 | 17 | 18 | 6 | 4
  Baseline: S2 | 147 | 14 | 19 | 3 | 9
  Baseline: S3 | 75 | 9 | 5 | 1 | 3
  Baseline: Missing | 3 | 0 | 0 | 0 | 0
  Month 6: number analyzed (Participants) | 302 | 72 | 50 | 15 | 20
  Month 6: S0 | 122 | 40 | 26 | 9 | 7
  Month 6: S1 | 70 | 19 | 15 | 3 | 9
  Month 6: S2 | 74 | 7 | 6 | 3 | 3
  Month 6: S3 | 32 | 5 | 3 | 0 | 1
  Month 6: Missing | 4 | 1 | 0 | 0 | 0
  Month 12: number analyzed (Participants) | 224 | 66 | 38 | 14 | 18
  Month 12: S0 | 110 | 39 | 25 | 10 | 6
  Month 12: S1 | 58 | 16 | 5 | 1 | 8
  Month 12: S2 | 40 | 6 | 5 | 2 | 4
  Month 12: S3 | 11 | 3 | 3 | 1 | 0
  Month 12: Missing | 5 | 2 | 0 | 0 | 0
  Month 18: number analyzed (Participants) | 168 | 53 | 32 | 8 | 17
  Month 18: S0 | 81 | 35 | 23 | 6 | 8
  Month 18: S1 | 41 | 11 | 5 | 0 | 4
  Month 18: S2 | 29 | 5 | 2 | 2 | 4
  Month 18: S3 | 15 | 1 | 2 | 0 | 1
  Month 18: Missing | 2 | 1 | 0 | 0 | 0
  Month 24: number analyzed (Participants) | 101 | 30 | 25 | 5 | 11
  Month 24: S0 | 71 | 20 | 17 | 3 | 7
  Month 24: S1 | 12 | 6 | 5 | 1 | 2
  Month 24: S2 | 12 | 3 | 1 | 1 | 2
  Month 24: S3 | 6 | 1 | 2 | 0 | 0
  Month 24: Missing | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Crohn's Disease: Number of Participants Categorized on the Basis of Fistula Drainage Assessment Index
Description: The fistula drainage assessment index was used to assess the improvement or remission of the disease activity of Crohn's Disease, based on 6 categories: remission (remission was defined as closure of all fistulae that were draining at baseline for at least two consecutive visits); improvement (improvement defined as a decrease from baseline in the number of open draining fistulae of 50% for at least two consecutive visits); worsened; unchanged; not accessible and missing disease activity.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 969 | 348 | 237 | 47 | 72
Participants
  Baseline: number analyzed (Participants) | 191 | 58 | 22 | 16 | 12
  Baseline: Remission | 64 | 30 | 14 | 3 | 6
  Baseline: Improvement | 90 | 26 | 5 | 11 | 4
  Baseline: Worsened | 9 | 0 | 0 | 0 | 0
  Baseline: Unchanged | 19 | 2 | 3 | 2 | 1
  Baseline: Not accessible | 4 | 0 | 0 | 0 | 1
  Baseline: Missing | 5 | 0 | 0 | 0 | 0
  Month 6: number analyzed (Participants) | 169 | 58 | 26 | 16 | 14
  Month 6: Remission | 65 | 29 | 17 | 6 | 8
  Month 6: Improvement | 62 | 23 | 3 | 9 | 4
  Month 6: Worsened | 12 | 1 | 3 | 1 | 0
  Month 6: Unchanged | 21 | 5 | 3 | 0 | 2
  Month 6: Not accessible | 4 | 0 | 0 | 0 | 0
  Month 6: Missing | 5 | 0 | 0 | 0 | 0
  Month 12: number analyzed (Participants) | 121 | 39 | 17 | 14 | 11
  Month 12: Remission | 50 | 23 | 11 | 9 | 9
  Month 12: Improvement | 39 | 8 | 3 | 1 | 0
  Month 12: Worsened | 9 | 0 | 0 | 1 | 0
  Month 12: Unchanged | 20 | 8 | 3 | 3 | 2
  Month 12: Not accessible | 1 | 0 | 0 | 0 | 0
  Month 12: Missing | 2 | 0 | 0 | 0 | 0
  Month 18: number analyzed (Participants) | 79 | 26 | 14 | 12 | 10
  Month 18: Remission | 36 | 16 | 9 | 6 | 8
  Month 18: Improvement | 23 | 4 | 1 | 2 | 0
  Month 18: Worsened | 5 | 1 | 0 | 2 | 0
  Month 18: Unchanged | 15 | 5 | 3 | 2 | 2
  Month 18: Not accessible | 0 | 0 | 1 | 0 | 0
  Month 18: Missing | 0 | 0 | 0 | 0 | 0
  Month 24: number analyzed (Participants) | 38 | 21 | 12 | 11 | 10
  Month 24: Remission | 16 | 12 | 4 | 7 | 7
  Month 24: Improvement | 8 | 6 | 3 | 3 | 1
  Month 24: Worsened | 3 | 0 | 2 | 0 | 0
  Month 24: Unchanged | 8 | 3 | 3 | 1 | 2
  Month 24: Not accessible | 1 | 0 | 0 | 0 | 0
  Month 24: Missing | 2 | 0 | 0 | 0 | 0

21. Secondary Outcome: Mean Change From Baseline in Laboratory Test Results: C-Reactive Protein at Months 6, 12, 18, and 24
Description: C-reactive protein (CRP) was a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultra-sensitive assay. A decrease in the level of CRP indicated reduction in inflammation and therefore improvement.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: FAS=all participants who received at least 1 dose of study drug and had at least one post-dose assessment of any of the effectiveness outcomes (clinical assessment of disease activity, laboratory and imaging results related to treatment or assessment of CD or UC). Here, Number analyzed =participants evaluable at specified time points for each arm.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1516 | 492 | 358 | 67 | 102
milligram per liter (mg/L)
  Baseline: number analyzed (Participants) | 1044 | 330 | 229 | 49 | 67
  Baseline | 13.70 (43.8) | 10.23 (22.6) | 8.79 (17.0) | 7.70 (11.8) | 12.18 (30.7)
  Change at Month 6: number analyzed (Participants) | 933 | 285 | 216 | 45 | 66
  Change at Month 6 | -1.09 (47.4) | 1.46 (40.0) | -1.45 (14.6) | -1.88 (12.3) | 0.94 (32.8)
  Change at Month 12: number analyzed (Participants) | 678 | 243 | 166 | 38 | 55
  Change at Month 12 | -4.87 (38.6) | -2.23 (17.3) | -1.62 (12.2) | 3.88 (25.4) | -4.84 (30.7)
  Change at Month 18: number analyzed (Participants) | 428 | 174 | 122 | 27 | 48
  Change at Month 18 | -6.57 (45.2) | 0.63 (37.7) | -2.45 (11.7) | 1.83 (12.6) | -0.59 (51.8)
  Change at Month 24: number analyzed (Participants) | 234 | 131 | 94 | 21 | 32
  Change at Month 24 | 0.33 (177.3) | -3.51 (18.2) | 3.19 (41.7) | 4.17 (24.6) | -3.11 (19.6)

22. Secondary Outcome: Mean Change From Baseline in Laboratory Test Results: Fecal Calprotectin at Months 6, 12, 18, and 24
Description: Here, the laboratory tests related to the treatment or assessment of Crohn's Disease or Ulcerative Colitis was fecal calprotectin.
Time Frame: Baseline, Months 6, 12, 18, and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: milligram per kilogram (mg/kg)
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1516 | 492 | 358 | 67 | 102
milligram per kilogram (mg/kg)
  Baseline: number analyzed (Participants) | 202 | 47 | 35 | 8 | 16
  Baseline | 1066.31 (5419.8) | 556.88 (916.2) | 362.48 (642.8) | 616.03 (1023.3) | 537.58 (1471.9)
  Change at Month 6: number analyzed (Participants) | 107 | 28 | 12 | 5 | 8
  Change at Month 6 | -283.21 (989.0) | -296.95 (958.1) | -164.60 (440.8) | -648.16 (1333.1) | 224.56 (700.1)
  Change at Month 12: number analyzed (Participants) | 55 | 22 | 10 | 2 | 7
  Change at Month 12 | -165.32 (691.9) | 361.51 (1741.1) | -289.57 (1004.9) | -382.73 (503.1) | -643.67 (2339.3)
  Change at Month 18: number analyzed (Participants) | 48 | 12 | 9 | 4 | 5
  Change at Month 18 | -473.07 (1394.3) | 275.48 (1518.0) | 88.44 (746.8) | -73.94 (125.3) | 109.16 (164.4)
  Change at Month 24: number analyzed (Participants) | 22 | 5 | 6 | 2 | 2
  Change at Month 24 | -625.69 (1684.7) | -862.40 (958.4) | -494.66 (1226.4) | -13.35 (273.4) | -450.98 (200.2)

23. Secondary Outcome: Number of Participants With Imaging Test Results
Description: Number of participants who had Imaging test results related to the treatment or assessment of Crohn's Disease or Ulcerative Colitis were reported.
Time Frame: From baseline up to follow-up period (a maximum of 2 years)
Population: FAS =all participants who received at least 1 dose of study drug and had at least one post-dose assessment of any of the effectiveness outcomes (clinical assessment of disease activity, laboratory and imaging results related to treatment or assessment of CD or UC).
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
Number analyzed (Participants) | 1516 | 492 | 358 | 67 | 102
Participants | 516 | 134 | 106 | 28 | 50

ADVERSE EVENTS:
Time Frame: From baseline to follow-up period (up to a maximum duration of 2 years)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population was evaluated.
Arm/Group | CT-P13 | Remicade | Switched From Remicade to CT-P13 | Switched From CT-P13 to Remicade | Multiple Switchers
All-Cause Mortality (participants affected / at risk) | 4/1522 | 2/494 | 1/358 | 0/67 | 0/102
Serious Adverse Events (participants affected / at risk) | 256/1522 | 43/494 | 57/358 | 10/67 | 15/102
Other Adverse Events (participants affected / at risk) | 442/1522 | 100/494 | 90/358 | 7/67 | 21/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P13 (N=1522) | Remicade (N=494) | Switched From Remicade to CT-P13 (N=358) | Switched From CT-P13 to Remicade (N=67) | Multiple Switchers (N=102)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 0 | 3 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 7 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 13 | 0 | 1 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 13 | 3 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 23 | 5 | 6 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal anastomotic stenosis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 11 | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 2 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 8 | 2 | 1 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 8 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Adhesion (General disorders) | 2 | 0 | 0 | 0 | 0
Administration site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0
Alcohol withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Condition aggravated (General disorders) | 1 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 11 | 1 | 5 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Paradoxical drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0
Stenosis (General disorders) | 0 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 1 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Lupus hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 5 | 0 | 0 | 2 | 1
Sarcoidosis (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Type I hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Abscess intestinal (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 5 | 1 | 3 | 0 | 0
Anal fistula infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Brain abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 4 | 0 | 0 | 0 | 1
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 2 | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected fistula (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Measles (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 0 | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 5 | 3 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
CSF pressure (Investigations) | 1 | 0 | 0 | 0 | 0
Drug specific antibody present (Investigations) | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Angiomyolipoma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle rupture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Meningioma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 3 | 2 | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Kidney congestion (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cervix carcinoma (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Caesarean section (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Colectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Behcet's syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Femoral artery embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P13 (N=1522) | Remicade (N=494) | Switched From Remicade to CT-P13 (N=358) | Switched From CT-P13 to Remicade (N=67) | Multiple Switchers (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 7 | 0 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal anastomotic stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Pouchitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 187 | 24 | 23 | 0 | 9
Dysplasia (General disorders) | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 1 | 4 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0
Fibrosis (General disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 0
Unevaluable event (General disorders) | 1 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 29 | 10 | 4 | 0 | 1
Serum sickness (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Type I hypersensitivity (Immune system disorders) | 9 | 2 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 5 | 2 | 1 | 0 | 0
Anal fistula infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 2 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Genital herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 4 | 0 | 3 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 3 | 2 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Opportunistic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Papilloma viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Parvovirus B19 infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pertussis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 4 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Ureteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 24 | 3 | 3 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 34 | 13 | 9 | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Suture related complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood count abnormal (Investigations) | 1 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Colonoscopy (Investigations) | 0 | 1 | 0 | 0 | 0
Drug specific antibody present (Investigations) | 6 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0
Mean cell volume decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 11 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Meningioma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 0 | 0
Gestational trophoblastic detachment (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 11 | 3 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Rebound psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 18 | 1 | 4 | 0 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Intestinal resection (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Poor venous access (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT02539368/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02539368/SAP_001.pdf